CLINICAL TRIAL: NCT00559065
Title: A Case - Cohort Study of Hematopoietic Malignancies and Related Disorders and Lung Cancer in Benzene-Exposed Workers in China
Brief Title: A Case-Cohort Study of Hematopoietic Malignancies and Related Disorders and Lung Cancer in Benzene-Exposed Workers in China
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: China for Disease Control (CDC) (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906205; 06-C-N205; NCT00516568 (obsolete NCT alias)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer; Lymphoma; Acute Non-Lymphocytic Leukemia; Benzene Poisoning; Leukemia
Keywords: Case-Cohort Study; Leukemia; Lymphoma; Benzene; Blood Disorders; Solvent Exposure; Cancer Risk
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Leukemia, Myeloid, Acute; Leukemia; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Benzene Cohort: Benzene exposed and unexposed workers.

SUMMARY:
This study will examine the risks of workplace exposure to benzene, a substance known to lead to cancer of the blood and possibly of the lungs. It is used widely in industries and is a contaminant in the environment. Researchers from the National Cancer Institute and the China Center for Disease Control (formerly Chinese Academy of Preventive Medicine) had done previous studies of workers in manufacturing industries in China of people who worked at least 1 day from 1972 to 1987 in 12 cities in that country. Data were collected of approximately 75,000 workers exposed to benzene and 35,000 who were not, with the purpose of investigating the relationship between benzene exposure and cancer risk. For workers exposed to benzene, there was a significant risk of cancer affecting the blood cells and a 1.8-fold excess of lung cancer among them. This study will expand those findings and also identify the effects of benzene amounts and whether there is a genetic tendency for benzene poisoning. About 3,860 benzene-exposed workers from the 12 cities will be interviewed. Next-of-kin of deceased workers, and a subcohort (additional grouping) of participants will serve as a control group in the research.

Patients who have worked at places where there was exposure to benzene will have a brief physical exam and samples of cells from a mouth rinse and samples from blood will be collected to study the genetic influence on developing blood diseases from workplace exposures.

All participants or next-of-kin, for deceased, will be given a questionnaire about their work history, use of cigarettes and hair dyes, medications they take, and family history of cancer. Interviews of about 40 minutes long will be conducted at participants homes or workplaces, at a time convenient to them, and the interviews will be audiotaped.

DETAILED DESCRIPTION:
Benzene is a known leukemogen and may cause lymphoma as well, but its ability to , cause these conditions below 10 parts per million (ppm) in air are unclear. It is currently regulated in the United States at 1 ppm as an 8-hour time-weighted average and at a 5 ppm short-term exposure level for 15 minutes. There is a critical need to assess risks related to benzene exposure under 10 ppm because it is widely used industrially and a ubiquitous contaminant in the environment.

The National Cancer Institute (NCI) and the Chinese Academy of Preventive Medicine (CAPM), whose name was recently changed to the China Center for Disease Control (CDC) previously established a cohort of 75,000 workers exposed to benzene in 12 cities in China and 35,000 unexposed comparison workers, to investigate the relationship between benzene exposure and cancer risk, from 1972 to 1987. We followed up each worker using factory records and reported results suggesting that benzene exposure under 10 ppm may be associated with increased risk of acute non-lymphocytic cancer and could also be associated with increased risk of lymphoma and lung cancer. We have now laid the groundwork for a further epidemiologic investigation in China to evaluate health risks from lower levels of benzene exposure, particularly as present in the factories during the 1990s. The cohort was followed up through 1999, and through this effort we have identified 3260 subjects for study, including cases (HLD malignancies, n= 161; benzene poisoning, n= 1040; lung cancer, n= 560) and 1500 subjects in a cohort sub-sample to be used as the comparison group. In addition, we have identified a series of cases with benzene poisoning and controls from the same factories outside of the cohort (n = 600).

We propose to contact next-of-kin of deceased subjects (essentially all cancer cases and some members of the sub-cohort are deceased), for questionnaire-based evaluation of benzene and other exposures, and to contact living subjects (primarily the benzene poisoning cases and the sub-cohort sample) for collection of questionnaires and biologic samples. The questionnaires (formatted for direct interview of living subjects or for next-of-kin) will collect information on potential confounders needed in the analysis of benzene's effects and information on work experience outside of the study cohort factories. The biologic sample collection (13 ml blood and buccal cell rinse) will provide material primarily for study of genetic polymorphisms potentially associated with benzene metabolism and disease status. The polymorphisms being studied are relatively common in the Chinese population and may be associated with a relatively modest increase in risk (1.5 to 2-fold). Written informed consent will be obtained from all next-of-kin and all live study subjects. We will attempt to enroll 3,860 study subjects or next-of-kin. The study will be carried out with Drs. Gui-Lan Li and Song-Nian Yin and colleagues from the China CDC, Beijing, China.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study subjects are Chinese. Gender is not an important consideration as a risk factor in benzene-exposed workers. Subjects will be recruited by on - site collaborators in each of the 12 study cities. Participation is voluntary. Subjects may withdra from the study at any time.

EXCLUSION CRITERIA:

Based on the available data, no cases (an , thus no controls) will be less than 18 years of age. Any subject under 18 would be excluded from the study. Otherwise, no exclusions of potential study subjects are planned.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From a cohort of 74,827 benzene-exposed and 35,804 unexposed workers employed (Bullet) one month in several industries and followed up during 1972-99, we identified a case-cohort population that included incident and deceased cases with hematopoietic malignancies diagnosed during those same years among exposed and unexposed workers and a 1,500 worker subcohort (1,100 exposed, 400 unexposed). The subcohort was selected by stratified random sampling (by sex, exposure status, and age at start of follow-up) from 106,641 of the cohort members. Other outcomes to be evaluated include incident cases with benzene hematotoxicity and deaths from lung cancer.
Sampling Method: Probability Sample
Enrollment: 3260 (Actual)
Dates: Start 2006-07-11 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Benzene poisoning, Hemapoietic Malignancies and related disorders, Lung cancer | 1972-1999
  Benzene poisoning, Hemapoietic Malignancies and related disorders, Lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Rothman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- China Center for Disease Control (CDC), Beijing, China

REFERENCES:
- [Background] Aksoy M. Malignancies due to occupational exposure to benzene. Am J Ind Med. 1985;7(5-6):395-402. doi: 10.1002/ajim.4700070506. PMID 4003402
- [Background] Aksoy M, Erdem S. Followup study on the mortality and the development of leukemia in 44 pancytopenic patients with chronic exposure to benzene. Blood. 1978 Aug;52(2):285-92. No abstract available. PMID 667356
- [Background] Arp EW Jr, Wolf PH, Checkoway H. Lymphocytic leukemia and exposures to benzene and other solvents in the rubber industry. J Occup Med. 1983 Aug;25(8):598-602. PMID 6886869